CLINICAL TRIAL: NCT05333250
Title: Modafinil to Improve Fatiguability (MODIFY): Modafinil vs. Placebo Vanguard RCT
Brief Title: Modafinil to Improve Fatiguability
Acronym: MODIFY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 663439
Record Dates: First submitted 2022-04-05; First posted 2022-04-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cancer-related Cognitive Difficulties; Cancer-related Problem/Condition; Fatigue
Keywords: Cancer; Fatigue; Cognitive Impairment; Modafinil
MeSH Terms: conditions — Fatigue; Neoplasms; Cognitive Dysfunction | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modafinil (Experimental): Two 100mg modafinil capsules once daily for 2 weeks
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Two 100mg placebo capsules once daily for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil
  Other Names: Provigil
  Arms: Modafinil
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Cancer-related fatigue (CRF) and cancer-related cognitive impairment (CRCI) are among the most commonly reported disabling symptoms experienced by patients with advanced cancer. However, there are currently limited evidence-based pharmacologic interventions available. The investigators will conduct a Vanguard Randomized Clinical Trial (RCT) to estimate the effect of modafinil in managing CRF and CRCI, and to test the feasibility of carrying out the study.

DETAILED DESCRIPTION:
Background:

Patients with advanced cancer often experience various disabling symptoms. Cancer-related fatigue (CRF) and cancer-related cognitive impairment (CRCI) are among the most common reported symptoms, yet the availability of evidence-based pharmacologic interventions is limited.

CRF can be defined as a "distressing, persistent, subjective sense of physical, emotional, and/or cognitive tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and interferes with usual functioning." CRF is experienced by over 75% of patients with advanced cancer.

CRCI is defined as a decline in one or more areas of cognitive function, including attention and concentration, executive functioning, information processing speed, language, visuospatial skill, psychomotor ability, and memory. It is estimated that up to 40% of patients experience CRCI prior to any treatment; up to 75% during their treatment; and up to 60% upon completion of therapies.

Modafinil is a psychostimulant that has been studied in the context of CRF and daytime sleepiness. Its mechanism of action is not clear, but it is thought to promote wakefulness through dopaminergic neurotransmission which has been hypothesized to play a role in CRF.

Study Hypothesis:

Modafinil will improve CRF and CRCI

Study Objectives:

1. To estimate the effect size of modafinil in managing CRF and CRCI
2. To test the feasibility of carrying out the study (recruitment, etc.)

Study Design:

Randomized, placebo-controlled, double-blind, single-centre vanguard trial

Sample Size & Study Population:

Approximately 40 outpatients presenting ≥4/10 on the fatigue score of their screening questionnaire will be recruited. Eligible patients must be 18-75 years old with advanced cancer who have not received cytotoxic chemotherapy for at least one month.

Intervention:

Subjects will be randomized to receive 200 mg of modafinil or placebo once daily for one week.

Study Outcome Measures:

Using validated questionnaires and a digital tool, the investigators will assess the patient's fatigue (CRF), cognition (CRCI), and quality of life before and after the intervention. In addition, patients will report their global impression of change.

Finally, if patients experience any adverse events (headache, nausea, vomiting, anxiety, etc.), they will report them using a standard questionnaire. Adverse events (AEs) and Serious Adverse Events (SAEs) will be documented.

Expected Outcomes:

Positive results should provide justification to prolong the study to complete a phase III trial. This study is important because fatigue remains a cause of suffering amongst palliative patients with cancer. Modafinil has the potential to improve patients' fatigue, cognition, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older with stage III or IV cancer diagnosis
2. Estimated prognosis ≥ 3 months
3. Eastern Cooperative Oncology Group (ECOG) Score 0-2
4. Experiencing cancer-related fatigue, defined as a score of 4 or greater on the Fatigue item of the Edmonton Symptom Assessment System-revised-constipation/sleep (ESAS-r-cs)
5. Ability to understand and communicate in English
6. Ability to give first-person informed consent

Exclusion Criteria:

* Currently receiving or have received cytotoxic chemotherapy in the last 6 weeks
* Allergy to modafinil or placebo contents
* Dose change of prednisone or dexamethasone in the past 7 days or planned dose change during study period
* Blood transfusion in the last 2 weeks
* Hemoglobin lower than 80 g/L measured in the last 4 weeks
* TSH above normal range in the last 4 weeks
* Severe liver dysfunction (total bilirubin >3x upper limit of normal, or aspartate aminotransferase or alanine aminotransferase >5x upper limit of normal)
* Known brain metastasis or primary brain tumor
* Documented dementia diagnosis
* Documented major psychiatric illness including major depressive episode, bipolar disorder, schizophrenia
* Uncontrolled hypertension as defined by a blood pressure greater than 140/90mmHg
* Unstable angina
* Recent (<6 months previous) myocardial infarction
* Evidence of left ventricular hypertrophy or ischemia on ECG
* Arrythmia (e.g., atrial fibrillation)
* Coronary artery disease with Canadian Cardiovascular Society Symptoms Class >1
* Taking high dose selective serotonin reuptake inhibitors (SSRIs) or tricyclic antidepressants
* Taking any benzodiazepine at any dose
* Taking any amphetamine at any dose
* Taking any monoamine oxidase inhibitor (MAOI) at any dose
* Taking any azole anti-fungal medication (e.g., fluconazole, itraconazole, or ketoconazole)
* Taking any of the following medications at any dose:

  1. Methylphenidate
  2. Cyclosporine
  3. Propranolol
  4. Phenytoin
  5. S-mephenytoin
  6. Warfarin
  7. Triazolam
  8. Ethinyl estradiol
  9. Clomipramine
  10. Midodrine
  11. Antipyrine
* Inability to ingest oral capsule
* Pregnancy or lactation, or trying to conceive
* Any other history, condition, therapy, or uncontrolled intercurrent illness which could, in the opinion of the Qualified Medical Investigator, affect compliance with study requirements or which would make the participant unsuitable for this study.
* Simultaneous participation in another interventional clinical study (e.g., Phase 1-3 clinical studies) or treatment with any investigational medicinal product within 30 days prior to screening visit that could, in the judgment of the Qualified Medical Investigator, affect the patient's participation in or outcome of this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 2 weeks
  Change in fatigue score evaluated using Multidimensional Fatigue Inventory (MFI).
Fatigue | 2 weeks
  Change in fatigue score evaluated using Patient's Global Impression of Change (PGIC) score.
Recruitment rate | 2 years
  The number of patients approached, total participants screened for eligibility, and reason for ineligibility or refusal to participate will be documented. We will consider the study successful if we can enroll 40 participants over a 2-year study period, with a recruitment rate of 15%.
Completion of intervention | 2 years
  We will consider the intervention to be feasible if at least 75% of enrolled participants complete the full intervention protocol.
Completion of follow-up | 2 years
  We will consider the intervention to be feasible if at least 75% of enrolled participants complete all assessments at 1-week follow-up.

SECONDARY OUTCOMES:
Cognition | 2 weeks
  Change in cognition score evaluated using the Fast Cognitive Evaluation (FaCE).
Quality of Life | 2 weeks
  Change in quality of life score evaluated using McGill Quality of Life Questionnaire-Revised (MQOL-R).
Adverse events | 2 weeks
  Daily patient-reported adverse effects with specific focus on headache, nausea and vomiting and anxiety, evaluated using the Common Terminology Criteria for Adverse Events (CTCAE).
Patient satisfaction with MFI | 2 weeks
  Patient satisfaction with MFI as a measure of their fatigue on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fitzgibbon, MD, MSc, CCFP(PC), Principal Investigator — The Ottawa Hospital; James Downar, MDCM, MHSc, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger AM, Mooney K, Alvarez-Perez A, Breitbart WS, Carpenter KM, Cella D, Cleeland C, Dotan E, Eisenberger MA, Escalante CP, Jacobsen PB, Jankowski C, LeBlanc T, Ligibel JA, Loggers ET, Mandrell B, Murphy BA, Palesh O, Pirl WF, Plaxe SC, Riba MB, Rugo HS, Salvador C, Wagner LI, Wagner-Johnston ND, Zachariah FJ, Bergman MA, Smith C; National comprehensive cancer network. Cancer-Related Fatigue, Version 2.2015. J Natl Compr Canc Netw. 2015 Aug;13(8):1012-39. doi: 10.6004/jnccn.2015.0122. PMID 26285247
- [Background] Jansen CE, Cancer Basics J, Eggert I (eds) (2010) Pittsburgh, PA:oncology nursing. Society
- [Background] Wefel JS, Kesler SR, Noll KR, Schagen SB. Clinical characteristics, pathophysiology, and management of noncentral nervous system cancer-related cognitive impairment in adults. CA Cancer J Clin. 2015 Mar;65(2):123-38. doi: 10.3322/caac.21258. Epub 2014 Dec 5. PMID 25483452
- [Background] Murillo-Rodriguez E, Barciela Veras A, Barbosa Rocha N, Budde H, Machado S. An Overview of the Clinical Uses, Pharmacology, and Safety of Modafinil. ACS Chem Neurosci. 2018 Feb 21;9(2):151-158. doi: 10.1021/acschemneuro.7b00374. Epub 2017 Dec 4. PMID 29115823
- [Background] Hovey E, de Souza P, Marx G, Parente P, Rapke T, Hill A, Bonaventura A, Michele A, Craft P, Abdi E, Lloyd A; MOTIF investigators. Phase III, randomized, double-blind, placebo-controlled study of modafinil for fatigue in patients treated with docetaxel-based chemotherapy. Support Care Cancer. 2014 May;22(5):1233-42. doi: 10.1007/s00520-013-2076-0. Epub 2013 Dec 17. PMID 24337761